CLINICAL TRIAL: NCT01558453
Title: Phase II Study With Oxaliplatin In Children With Relapsed/Refractory Solid Tumors
Brief Title: Oxaliplatin for Children With Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sidnei Epelman (Other)
Responsible Party: Sponsor-Investigator, Sidnei Epelman, Director of Pediatric Oncology Department, Hospital Santa Marcelina
Organization: Hospital Santa Marcelina (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_04946
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Relapsed Solid Tumor; Refractory Solid Tumor
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eloxatin (Experimental): Oxaliplatin
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered in a 130 mg/m² dose, 2 hour IV infusion, once every 3 weeks. Each cycle will last 3 weeks, or 21 days. Drug will be administered till progression disease or untolerable adverse event.
  NOTE: patients with ≤ 12 months old will receive a 4,3 mg/kg dese (based on a 30 kg/m² conversion; i.e: in a 130 mg/m² dose, divided by 30).

SUMMARY:
The purpose of this study is to determine the pediatric neoplastic response to chemotherapy proposed and evaluate sensitivity to oxaliplatin through immunohistochemistry ERCC-1 expression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 21 years old at the time of cancer diagnosis.
2. Confirmed histological diagnosis - every patient, except brains tumor, or optic pathway glioma, should have one of the following histological diagnosis:

   * Ewing´s sarcoma/PNET
   * Osteosarcoma
   * Soft tissue sarcoma/rhabdomyosarcoma
   * Wilms tumor
   * Neuroblastoma
   * Retinoblastoma
   * Low grade astrocytoma
   * High grade astrocytoma/GBM
   * Ependymoma
   * Germ cell tumor Other rare tumors such as - hepatocellular carcinoma, pediatric colorectal carcinoma, renal cell carcinoma, adrenocortical carcinoma and nasopharyngeal carcinoma.
3. All subjects should have measurable disease, at least in one dimension, 20mm minimum, or presence of neoplastic cell in cephalorachidian fluid.
4. All patients must have a life expectancy ≥ 8 weeks, with PS Karnofsky ≥50 for patients with ≥ 10 years old and PS Lansky ≥50 for patients < 10 years old.
5. Previous treatment:

   * at least 3 weeks without chemotherapy.
   * at least 6 months after spine and brain radiation.
   * it is allowed corticosteroids in patients with CNS tumor, but it is recommended to have stable doses or reducing the dose 7 days before protocol treatment.
   * there´s no limit of drugs or chemotherapy used previously, except oxaliplatin.
6. Adequate function as define by:

   * Hematologic: neutrophil > 1000/mm³, platelet > 75000/mm³ and hemoglobin > 8 g/dL.
   * Renal - creatinine according to:

   Age ≤ 5 anos Cr ≤ 0,8 mg/dL 5 < age < 10 Cr ≤ 1,0 mg/dL 10 < age ≤ 15 Cr ≤ 1,2 mg/dL > 15 years Cr ≤ 1,5 mg/dL
   * Hepatic: total bilirubin ≤ 3 mg/dL.
   * Neurologic: patients should seizure control.
7. Legal representative (father, mother or tutor) or subject (if >18 years old) must sign and date Informed Consent Form (ICF), after have being informed about relevant aspects regarding study participation.
8. For female patients of childbearing age: Presence of a negative pregnancy test within 7 days prior to day 0.
9. Patient must agree in use effective contraception if procreative potential exists. Use of reliable means of contraception (e.g. hormonal contraceptive, patch, vaginal ring, intrauterine device, physical barrier, abstinence) for subjects of reproductive potential (males and females) is required during study treatment and for 3 months following last dose of study drug
10. It should not have known curative treatment option and no proved therapy that increased survival with quality of life.

Exclusion Criteria:

1. Oxaliplatin previous use.
2. Another chemotherapy or experimental drug, simultaneously.
3. If female, pregnant or lactating.
4. Active infection.
5. Any serious existent condition that could affect, in adverse way, subjet's capacity to be treat according to protocol.
6. Any condition, therapy, or medical condition, which, in the opinion of the attending physician could represent a risk for the patient or adversely affect the study objectives.
7. Use of investigational drug < 30 days before entering study.
8. Medical history with:

   * severe renal insufficiency;
   * known hypersensitiveness to platine;
   * myelosuppression;
   * peripheral sensory neuropathy.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determine pediatric neoplastic response to proposed chemotherapy. Evaluate sensitivity to oxaliplatin through immunohistochemistry ERCC-1 expression analysis. | Up 2 years

SECONDARY OUTCOMES:
Define cumulative toxicity after oxaliplatin multiple cycles in this population. Evaluate relation between time exposure to the drug (number of cycles) and response (antitumor effect x response). | Up 2 years
  Determine response time and overall survival in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sidnei Epelman, MD, Study Chair — Santa Marcelina Hospital
Locations (1):
- Santa Marcelina Hospital, São Paulo, São Paulo, Brazil